CLINICAL TRIAL: NCT00650858
Title: Clot Lysis: Evaluating Accelerated Resolution of Intraventricular Hemorrhage (IVH)
Brief Title: Clinical Trial on Treatment of Intraventricular Hemorrhage
Acronym: CLEAR IVH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: FDA Office of Orphan Products Development (U.S. Federal Agency); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IVH05; ISRCTN47341677 (Registry Identifier: ISRCTN registry)
Record Dates: First submitted 2007-12-26; First posted 2008-04-02 (Estimated); Results first posted 2012-07-17 (Estimated); Last update posted 2017-12-11 (Actual); Status verified 2017-11

CONDITIONS: Intraventricular Hemorrhage
Keywords: Intraventricular hemorrhage (IVH); rt-PA
MeSH Terms: interventions — Tissue Plasminogen Activator; Fibrinolytic Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 0.3 mg rt-PA (Active Comparator): In stage 1 of the protocol, dose finding, subjects were randomized to either this 0.3 mg dose arm or the 1.0 mg dose arm. Subjects in this arm (0.3 mg) received up to 8 doses of 0.3 mg rt-PA every 12 hours through the intraventricular catheter to treat intraventricular hemorrhage.
  Interventions: Drug: tissue plasminogen activator, rt-PA (thrombolytic) (Cathflo)
- 1.0 mg rt-PA (Active Comparator): In stage 1 of the protocol, dose finding, subjects were randomized to either this 1.0 mg dose arm or the 0.3 mg dose arm. Subjects in this arm (1.0 mg) received up to 8 doses of 1.0 mg rt-PA every 12 hours through the intraventricular catheter to treat intraventricular hemorrhage.
  Interventions: Drug: tissue plasminogen activator, rt-PA (thrombolytic) (Cathflo)
- 1.0 mg Rt-PA q8h (Experimental): In stage 2 of the protocol, dose frequency, subjects received up to 8 doses of 1.0 mg of rt-PA (Cathflo) every 8 hours through the intraventricular catheter to treat intraventricular hemorrhage.
  Interventions: Drug: tissue plasminogen activator, rt-PA (thrombolytic) (Cathflo)

INTERVENTIONS:
Drug: tissue plasminogen activator, rt-PA (thrombolytic) (Cathflo) — 0.3 mg and 1.0 mg of rt-PA (Cathflo) were administered every 12 hours (dose finding) and every 8 hours (dose frequency) via the intraventricular catheter to treat intraventricular hemorrhage.
  Other Names: rt-PA; Cathflo; Activase

SUMMARY:
The specific objective of this trial is to determine the lowest dose and dose frequency possible with the best pharmacokinetic and safety profile and it's ability to remove a blood clot from the ventricular system.

DETAILED DESCRIPTION:
The purpose of this trial is to determine the efficacy and pharmacokinetics of intraventricular injections of multiple low doses of rt-PA. Sixteen subjects were already randomized to receive intraventricular injections of with 0.3 mg or 1.0 mg of rt-PA every 12 hours for up to 8 doses. Results of this stage (n=16) were then analyzed and the most effective dose of 1.0 mg was chosen to be used in the second stage (n=36) to determine the optimal frequency of dosing. We propose to test if this intervention facilitates more rapid clot resolution, complete recovery function and decreased mortality from this condition.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75
2. IVC placed as standard of care using less than or equal to 2 complete passes.
3. Spontaneous ICH less than or equal to 30 cc.
4. Able to receive first dose within 48 hours of CT scan diagnosing IVH (providing the time of symptom onset to diagnostic CT does not exceed 12 hours).
5. Clot size measured on CT scan done 6 hours after IVC placement must be equal to the presentation clot size plus or minus 5 cc (as determined by the AxBxC)/2 method).
6. ON stability CT scan either the 3rd or 4th ventricles are occluded with blood (no evidence of CSF flow on CT).
7. SBP < 200 mmHg sustained for 6 hours.
8. Historical Rankin of 0 or 1.

Exclusion Criteria:

1. Suspected or untreated aneurysm or AVM (unless ruled out by angiogram or MRA/MRI).
2. Clotting disorders.
3. Patients with platelet count < 100,000, INR > 1.7, PT > 15s, or an elevated APTT.
4. Pregnancy (positive pregnancy test).
5. Infratentorial hemorrhage (i.e., parenchymal/posterior fossa hematoma; all cerebellar hematomas excluded).
6. SAH (An angiogram should be obtained when the diagnostic CT scan demonstrates subarachnoid hemorrhage or any hematoma location or appearance not strongly associated with hypertension. If the angiogram does not demonstrate a bleeding source that accounts for the hemorrhage, the patient is eligible for the study).
7. ICH enlargement during the 6-hour stabilization period (6 hour after IVC placement).
8. Internal bleeding, involving retroperitoneal sites, or the gastrointestinal, genitourinary, or respiratory tracts.
9. Superficial or surface bleeding, observed mainly at vascular puncture and access sites (e.g., venous cutdowns, arterial punctures) or site of recent surgical intervention.
10. Known risk for embolization, including history of left heart thrombus, mitral stenosis with atrial fibrillation, acute pericarditis, and subacute bacterial endocarditis.
11. Prior enrollment in the study.
12. Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated.
13. Participation in another simultaneous medical investigation or trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2004-02; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel F Hanley, MD, Study Chair — Johns Hopkins University
Locations (25):
- United States (22):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - CR Drew Medical Center, Los Angeles, California
  - Standford Medical Center, Palo Alto, California
  - Hartford Hospital, Hartford, Connecticut
  - Loyola University Medical Center, Maywood, Illinois
  - Via Christi Regional Medical Center, Wichita, Kansas
  - University of Maryland Medical Systems, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Wayne State University, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - St. Louis University, St Louis, Missouri
  - Albany Medical Center, Albany, New York
  - Mt. Sinai Medical Center, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Temple University, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor College of Medicine, Houston, Texas
  - University of Texas HSC, San Antonio, San Antonio, Texas
  - University of Virginia, Charlottesville, Charlottesville, Virginia
  - INOVA Fairfax Medical Center, Fairfax, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Foothills Medical Centre, Calgary, Alberta, Canada
- University of Heidelberg, Heidelberg, Germany
- Newcastle General Hospital, Newcastle upon Tyne, United Kingdom

REFERENCES:
- [Derived] Kornbluth J, Nekoovaght-Tak S, Ullman N, Carhuapoma JR, Hanley DF, Ziai W. Early Quantification of Hematoma Hounsfield Units on Noncontrast CT in Acute Intraventricular Hemorrhage Predicts Ventricular Clearance after Intraventricular Thrombolysis. AJNR Am J Neuroradiol. 2015 Sep;36(9):1609-15. doi: 10.3174/ajnr.A4393. Epub 2015 Jul 30. PMID 26228884
- [Derived] Ziai W, Moullaali T, Nekoovaght-Tak S, Ullman N, Brooks JS, Morgan TC, Hanley DF. No exacerbation of perihematomal edema with intraventricular tissue plasminogen activator in patients with spontaneous intraventricular hemorrhage. Neurocrit Care. 2013 Jun;18(3):354-61. doi: 10.1007/s12028-013-9826-1. PMID 23463422
- [Derived] Morgan TC, Dawson J, Spengler D, Lees KR, Aldrich C, Mishra NK, Lane K, Quinn TJ, Diener-West M, Weir CJ, Higgins P, Rafferty M, Kinsley K, Ziai W, Awad I, Walters MR, Hanley D; CLEAR and VISTA Investigators. The Modified Graeb Score: an enhanced tool for intraventricular hemorrhage measurement and prediction of functional outcome. Stroke. 2013 Mar;44(3):635-41. doi: 10.1161/STROKEAHA.112.670653. Epub 2013 Jan 31. PMID 23370203
- [Derived] Webb AJ, Ullman NL, Mann S, Muschelli J, Awad IA, Hanley DF. Resolution of intraventricular hemorrhage varies by ventricular region and dose of intraventricular thrombolytic: the Clot Lysis: Evaluating Accelerated Resolution of IVH (CLEAR IVH) program. Stroke. 2012 Jun;43(6):1666-8. doi: 10.1161/STROKEAHA.112.650523. Epub 2012 Apr 3. PMID 22474059
- [Derived] Ziai WC, Muschelli J, Thompson CB, Keyl PM, Lane K, Shao S, Hanley DF. Factors affecting clot lysis rates in patients with spontaneous intraventricular hemorrhage. Stroke. 2012 May;43(5):1234-9. doi: 10.1161/STROKEAHA.111.641050. Epub 2012 Mar 1. PMID 22382155
- [Derived] Herrick DB, Ziai WC, Thompson CB, Lane K, McBee NA, Hanley DF. Systemic hematologic status following intraventricular recombinant tissue-type plasminogen activator for intraventricular hemorrhage: the CLEAR IVH Study Group. Stroke. 2011 Dec;42(12):3631-3. doi: 10.1161/STROKEAHA.111.625749. Epub 2011 Sep 22. PMID 21940973
- See also: CLEAR III Website — http://www.cleariii.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began for protocol stage 1 in August 2005 and ended for protocol stage 2 on February 6, 2008. Subjects were screened by clinical stroke service personnel in the Emergency Department or by direct transfer from an outside hospital.
Groups:
- 0.3 mg Rt-PA q12h; 1.0 mg Rt-PA q12h: Stage 1 (Dose Finding)
- 1.0 mg Rt-PA q8h: Stage 2 (Dose Optimization)
Period: Overall Study
Arm/Group | 0.3 mg Rt-PA q12h | 1.0 mg Rt-PA q12h | 1.0 mg Rt-PA q8h
Started | 8 | 8 | 36
Completed | 8 | 8 | 36
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.3 mg Rt-PA q12h | 1.0 mg Rt-PA q12h | 1.0 mg Rt-PA q8h | Total
Number analyzed (Participants) | 8 | 8 | 36 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 26 | 39
  >=65 years | 1 | 2 | 10 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.6 (9.8) | 57.3 (8.3) | 57.0 (10.2) | 55.6 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 11 | 18
  Male | 5 | 4 | 25 | 34
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 31 | 47
  Canada | 0 | 0 | 3 | 3
  Germany | 0 | 0 | 1 | 1
  United Kingdom | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: 30-day Mortality
Description: The number of subjects who died at or before the 30-day follow-up visit were determined as a measure of safety. If more than 50% of the subjects died at or before the 30-day follow-up visit, the study would have been stopped for full DSMB review.
Time Frame: 30 days
Measure: Number; unit: Number of participants
Arm/Group | 0.3 mg Rt-PA q12h | 1.0 mg Rt-PA q12h | 1.0 mg Rt-PA q8h
Number analyzed (Participants) | 8 | 8 | 36
Number of participants | 1 | 1 | 6

2. Primary Outcome: Incidence of Bacterial Ventriculitis, Meningitis
Description: The incidence of bacterial ventriculitis/meningitis was recorded to determine the safety of intraventricular administration of rt-PA. If 30% or more subjects experienced this event, the study would have been stopped for full DSMB review.
Time Frame: 30 days
Measure: Number; unit: Number of participants
Arm/Group | 0.3 mg Rt-PA q12h | 1.0 mg Rt-PA q12h | 1.0 mg Rt-PA q8h
Number analyzed (Participants) | 8 | 8 | 36
Number of participants | 0 | 1 | 1

3. Primary Outcome: Rate of Symptomatic Bleeding Events
Description: The rate of symptomatic brain bleeding events were recorded to determine the safety of intraventricular administrations of rt-PA. If 35% or more subjects experienced a symptomatic bleeding event prior to the 30-day follow-up visit, the study would have been stopped for a full DSMB review.
Time Frame: 30-days
Measure: Number; unit: participants
Arm/Group | 0.3 mg Rt-PA q12h | 1.0 mg Rt-PA q12h | 1.0 mg Rt-PA q8h
Number analyzed (Participants) | 8 | 8 | 36
participants | 0 | 0 | 2

4. Secondary Outcome: Average Daily Percentage Clot Size Resolution Over the First 3 Days
Description: Daily IVH clot volume resolution, as a percentage of stability CT IVH volume, averaged over the first 3 days, determined by CT scans
Time Frame: 3 days
Measure: Mean (Full Range); unit: Percent of stability CT volume resolved
Arm/Group | 0.3 mg Rt-PA q12h | 1.0 mg Rt-PA q12h | 1.0 mg Rt-PA q8h
Number analyzed (Participants) | 8 | 8 | 36
Percent of stability CT volume resolved | 22.19 [8 to 66] | 24.20 [0 to 72] | 19.99 [0 to 60]

5. Secondary Outcome: 90 Day Follow-Up Modified Rankin Scale (mRS) Score
Description: 90 day follow-up visit mRS score. The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. It is scored from 0 to 6: 0. No Symptoms, 1. No Significant Disability, 2. Slight Disability, 3. Moderate Disability, 4. Moderately Severe Disability, 5. Severe Disability and 6. Dead.
  (Stage 1 patients only had 30 day scores, Stage 2 patients had 30 day, 90 day and 180 day scores collected)
Time Frame: 90 days
Measure: Median (Full Range); unit: mRS score
Arm/Group | 0.3 mg Rt-PA q12h | 1.0 mg Rt-PA q12h | 1.0 mg Rt-PA q8h
Number analyzed (Participants) | 0 | 0 | 36
mRS score |  |  | 4.3 [0 to 6]

6. Secondary Outcome: 90 Day Follow-Up Glasgow Outcome Scale (GOS) Score
Description: 90 day follow-up visit GOS score. The GOS is a scale used to determine the degree of recovery from patients with brain injury. There are five categories: 1. Dead, 2. Vegetative State, 3. Severe Disability, 4. Moderate Disability and 5. Good Recovery.
  (Stage 1 patients only had 30 day scores, Stage 2 patients had 30 day, 90 day and 180 day scores collected)
Time Frame: 90 days
Measure: Median (Full Range); unit: GOS score
Arm/Group | 0.3 mg Rt-PA q12h | 1.0 mg Rt-PA q12h | 1.0 mg Rt-PA q8h
Number analyzed (Participants) | 0 | 0 | 35
GOS score |  |  | 2.3 [0 to 4]

7. Secondary Outcome: 180 Day Follow-Up Modified Rankin Scale (mRS) Score
Description: 180 day follow-up visit mRS score. The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. It is scored from 0 to 6: 0. No Symptoms, 1. No Significant Disability, 2. Slight Disability, 3. Moderate Disability, 4. Moderately Severe Disability, 5. Severe Disability and 6. Dead.
  (Stage 1 patients only had 30 day scores, Stage 2 patients had 30 day, 90 day and 180 day scores collected)
Time Frame: 180 days
Measure: Median (Full Range); unit: mRS score
Arm/Group | 0.3 mg Rt-PA q12h | 1.0 mg Rt-PA q12h | 1.0 mg Rt-PA q8h
Number analyzed (Participants) | 0 | 0 | 35
mRS score |  |  | 4.0 [0 to 6]

8. Secondary Outcome: 180 Day Follow-Up Glasgow Outcome Scale (GOS) Score
Description: 180 day follow-up visit GOS score. The GOS is a scale used to determine the degree of recovery from patients with brain injury. There are five categories: 1. Dead, 2. Vegetative State, 3. Severe Disability, 4. Moderate Disability and 5. Good Recovery.
  (Stage 1 patients only had 30 day scores, Stage 2 patients had 30 day, 90 day and 180 day scores collected)
Time Frame: 180 days
Measure: Median (Full Range); unit: GOS score
Arm/Group | 0.3 mg Rt-PA q12h | 1.0 mg Rt-PA q12h | 1.0 mg Rt-PA q8h
Number analyzed (Participants) | 0 | 0 | 35
GOS score |  |  | 2.3 [0 to 4]

ADVERSE EVENTS:
Arm/Group | 0.3 mg Rt-PA q12h | 1.0 mg Rt-PA q12h | 1.0 mg Rt-PA q8h
Serious Adverse Events (participants affected / at risk) | 3/8 | 2/8 | 11/36
Other Adverse Events (participants affected / at risk) | 7/8 | 8/8 | 32/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.3 mg Rt-PA q12h (N=8) | 1.0 mg Rt-PA q12h (N=8) | 1.0 mg Rt-PA q8h (N=36)
Accidental Extubation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0) | 3 (3)
Cerebral Infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hemorrhage new catheter tract >5 mm with mass effect, symptomatic (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hydrocephalus, Communicating (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
ICH Hemorrhage, new symptomatic (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
IVH Hemorrhage enlargement - asymptomatic (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
IVH Hemorrhage enlargement - symptomatic (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
IVH hemorrhage, new symptomatic (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Suspected cardiac or pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Tracheal stricture (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ventilatory failure, mechanical (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Ventriculitis, Bacterial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Ventriculitis, non-bacterial (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.3 mg Rt-PA q12h (N=8) | 1.0 mg Rt-PA q12h (N=8) | 1.0 mg Rt-PA q8h (N=36)
Acute Renal Failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Adult Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2)
Bacteremia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (4)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Brain Edema / Swelling (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3)
CSF Leak (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Cerebral Infarction (Nervous system disorders) | 0 (0) | 0 (0) | 5 (5)
Cerebral infarction, extension (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Congestive Heart Failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Decreased Level of counciousness (Nervous system disorders) | 3 (3) | 2 (2) | 7 (12)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3)
Edema (metabolic causes) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Fever of unknown origin (General disorders) | 3 (3) | 4 (4) | 8 (8)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 3 (4)
Hemorrhage enl, cath tract >5mm w/o mass, asym (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2)
Hemorrhage enlargement, catheter tract > 5 mm with mass effect, asymptomatic (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Hemorrhage, new catheter tract <= 5 mm, asymptomatic (Nervous system disorders) | 0 (0) | 3 (3) | 2 (2)
Hemorrhage, new catheter tract > 5 mm with mass effect, asymptomatic (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Hemorrhage, new catheter tract > 5 mm with mass effect, symptomatic (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Herniation, Brain (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hydrocephalus, Obstructive (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hydrocephalus, communicating (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3)
Hyperglycemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Cardiac disorders) | 1 (1) | 3 (4) | 1 (1)
Hypokalemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 3 (3)
Hyponatremia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Hypoxemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
ICH hemorrhage enlargement, asymptomatic (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
ICH hemorrhage, new asymptomatic (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
ICH hemorrhage, new symptomatic (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
IVH hemorrhage enlargement - asymptomatic (Nervous system disorders) | 0 (0) | 0 (0) | 3 (4)
Increased Blood Urea Nitrogen (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Increased midline shift (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Intracranial hypertension (Nervous system disorders) | 1 (5) | 2 (2) | 2 (4)
Peri-hemorrhagic ischemic change (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 9 (9)
Pneumonia, aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (3)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
SAH Hemorrhage, new asymptomatic (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Siezure (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Skin Exanthema (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tracheitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 2 (2) | 4 (4)
Ventilatory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Ventriculitis, bacterial (Nervous system disorders) | 0 (0) | 1 (1) | 2 (4)
Ventriculitis, non-bacterial (Nervous system disorders) | 0 (0) | 1 (1) | 8 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI shall provide the sponsor with a copy of any proposed publication for review and comment thirty (30) days prior to submission. JHU may request a delay in publication, not to exceed 90 days if it is necessary to protect any intellectual property.